CLINICAL TRIAL: NCT07006636
Title: Effect of Watermelon Consumption on Cardiometabolic Health and Whole-Body Antioxidant Capacity
Brief Title: Effect of Watermelon on Cardiometabolic Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Watermelon Promotion Board (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-25-1126
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-08

CONDITIONS: Cardiometabolic Health Indicators; Whole-body Antioxidant Capacity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Watermelon Juice + liquid meal test at baseline (Experimental): Acute (postprandial) as well as chronic (4 weeks) effects of WMJ consumption will be evaluated. To evaluate acute effects participants will consume a liquid meal test together with WMJ at the beginning of the intervention phase. In addition, the same liquid meal test will be consumed with only WMJ at the end of the intervention phase to assess whether drinking the juice for 4 weeks prior had any effects on postprandial responses.
  Interventions: Other: Watermelon Juice + liquid meal test at baseline
- Sweetened placebo beverage + liquid meal test at baseline (Placebo Comparator): Participants will consume placebo beverage + liquid meal test at baseline. They will then consume watermelon juice daily for 4 weeks. Watermelon juice + liquid meal test will be consumed at endpoint.
  Interventions: Other: Sweetened placebo beverage +liquid meal test at baseline

INTERVENTIONS:
Other: Watermelon Juice + liquid meal test at baseline — WMJ will be purchased from a commercially available brand. The liquid meal test will be in the form of the Boost nutritional drink (8 fl.oz., vanilla flavor), which is commercially available.
  Arms: Watermelon Juice + liquid meal test at baseline
Other: Sweetened placebo beverage +liquid meal test at baseline — The placebo beverage made of water and sugar will match the sugar content provided in 355 ml of WMJ (approximately 10-20 g). The liquid meal test will be in the form of the Boost nutritional drink (8 fl.oz., vanilla flavor), which is commercially available.
  Arms: Sweetened placebo beverage + liquid meal test at baseline

SUMMARY:
The purpose of this study is to determine whether consumption of 355 ml of watermelon juice will:

1. improve cardiovascular and overall metabolic health markers like blood pressure, heart rate, stiffness/flexibility of arteries (blood vessels), blood sugar, cholesterol), and gut hormones
2. contribute to the body's ability to protect itself from the potential cell damage caused by harmful chemical compounds (produced when skin is exposed to ultraviolet (UV) B light, for example). This will be evaluated by measuring how resistant skin is to the damage from UVB light exposure, as well as several markers of bodily stress blood and urine.

This will be determined immediately after consuming the juice (to evaluate the effects the juice has on health right away), as well as after 4 weeks of daily juice consumption (to evaluate the effects the juice has on health when consumed consistently over time).

DETAILED DESCRIPTION:
Both hypertension and oxidative stress are among the major risk factors for cardiovascular disease (CVD). While CVD is a multifactorial disease, it has been established that diet plays an integral role in its pathogenesis. In fact, it has been previously demonstrated that almond and pomegranate consumption may be able to strengthen the body's antioxidant defense mechanisms and aid in improving several cardiometabolic health biomarkers. Watermelon, being rich in fiber, vitamins, minerals, and bioactive compounds (e.g., L-citrulline, lycopene, beta-carotene) may also have similar health effects. Notably, studies involving both mice and humans have demonstrated the potential of watermelon consumption to prevent CVD by lowering blood pressure and low-density lipoprotein cholesterol (LDL-C).

Emerging evidence suggests that postprandial biomarker levels may serve as better and earlier predictors of CVD development than their fasting levels. While watermelon is often consumed with or after a meal, no studies have evaluated the effect of watermelon on postprandial biomarker responses after a meal challenge. In addition, despite the high bioactive content of watermelon, its effects on whole-body antioxidant capacity have not been explored yet.

Therefore, in the present study it is proposed to evaluate the acute (postprandial) and chronic (4 weeks of daily consumption) effects of 355 ml of watermelon juice (WMJ) on: 1) cardiometabolic risk factors including blood pressure, heart rate, pulse wave velocity (PWV), blood glucose and lipids/lipoproteins, nitric oxide (NO), insulin/C-peptide, and GLP-1; and 2) whole-body antioxidant capacity by evaluating skin resistance to UV irritation, as well as blood and urine malondialdehyde (MDA) levels. A two-phase intervention study (2-week standardization phase and a 4-week intervention phase) involving 20 generally healthy non-vegetarian/vegan postmenopausal women with slightly elevated blood pressure, overweight/obese BMI, and Fitzpatrick's skin types II-IV will be performed. Investigating the effects of WMJ consumption on cardiometabolic risk factors and skin antioxidant defense/systemic oxidative status will uncover valuable new insights into whether bioactive compounds in watermelon can affect cardiometabolic risk and contribute to the total body antioxidant capacity.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Generally healthy
* Postmenopausal
* BMI 25-40 kg/m2
* Systolic blood pressure 120-139 mmHg and/or diastolic 80-89 mmHg
* Fitzpatrick Skin type II-IV
* Consume a typical Western diet (low in polyphenol/lycopene-rich foods and fiber)
* Willing to maintain habitual dietary and exercise patterns for the study duration
* Willing to maintain normal skin care products and pattern for the duration of the study
* Willing to come to Baseline Visit B and Week 4 study visits without any makeup and skin products on
* Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent.

Exclusion Criteria:

* Non-English speaker
* Vegetarian/vegan
* Known watermelon allergy
* Skin-related prescription medication, supplements, or non-prescription cosmeceutical agents
* Initiation of topical or oral prescription steroids and/or anti-inflammatory medications within 30 days prior to study enrollment
* Excessive exposure to either natural or artificial sunlight. Exposure to sunlight will be evaluated using Fitzpatrick Skin Type test score. Individuals receiving scores higher than the upper cutoff of the proposed range for the specific skin type will be excluded
* Screening laboratory values outside of the normal range that is considered clinically significant for study participation by the investigator
* Documented chronic disease, including diabetes, renal or liver diseases, metabolic syndrome, active cancer, MI or stroke, history of gastric bypass or GI disease (e.g., Crohn's disease, IBD, diverticulosis, diverticulitis, etc.)
* Taking medications or supplements known to affect metabolism or gut microbiota composition (antibiotics within the past 3 months, probiotics, fiber, etc.), unless willing to stop for the study duration
* Taking exogenous hormones (e.g., hormone replacement therapy)
* Recent weight fluctuations (>10% in the last 6 months)
* Smoker or living with a smoker
* Use of >20 g of alcohol per day
* Unable or unwilling to comply with the study protocol (including unwillingness to avoid watermelon and other lycopene-rich foods for the whole duration of the study)
* Unable to provide consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Postprandial blood pressure | Baseline and Week 4
  To determine the acute and chronic effects of WMJ consumption on cardiometabolic health, specifically focusing on postprandial blood pressure. Previous studies showed that watermelon extract improved blood pressure management in subjects with prehypertension and hypertension and reduced arterial stiffness in postmenopausal women. Postprandial blood pressure response is recently identified to be the most sensitive postprandial clinical feature in predicting subclinical atherosclerosis. However, no study has evaluated the effect of watermelon on postprandial blood pressure. Blood pressure will be measured in mm/Hg.
Postprandial heart rate | Baseline and 4 weeks.
  Will be measured in beats per minute.
Postprandial pulse wave velocity | Baseline and 4 weeks.
  Will be measured in meters/second.

SECONDARY OUTCOMES:
Postprandial nitric oxide (NO) | Baseline and 4 weeks.
  Will be measured in µmol/L
Postprandial glucose | Baseline and 4 weeks.
  Dysregulation of postprandial glucose and lipid responses has been implicated in the development of metabolic diseases. A previous study showed that watermelon juice consumption acutely stabilized postprandial glucose and insulin levels compared to matched sugar water in healthy subjects. Here, we will evaluate both acute and chronic effects of watermelon juice on postprandial circulating biomarker responses.
Postprandial blood lipids/lipoproteins (LDL cholesterol, HDL cholesterol, total cholesterol, triglycerides). | Baseline and 4 weeks.
  All will be measured in mg/dL.
Postprandial insulin | Baseline and 4 weeks.
  Will be measured in international units.
Postprandial C-peptide | Baseline and 4 weeks.
  Will be measured in nmol/L
Postprandial GLP-1 | Baseline and week 4
  Will be measured in pmol/L

OTHER OUTCOMES:
Minimal Erythema Dose (MED) | Baseline and week 4.
  Based on overall skin type classification, we will use the National Biological UVB mJ chart to determine the dose and sequential exposure times. Using the SPF Solar Simulator (Solar light, PA), participants' inner arm will be irradiated with a defined dose of UVB light. A total of six gradually increasing doses will be used. The subjects will return 24 hours later to determine which skin area shows minimal erythema (pink color). Photographs will be taken before irradiation and after 24 hours. The lowest dose and time of the occurrence of pink will be determined and used as MED.
Blood and urinary malondialdehyde (MDA) concentrations | Baseline and 4 weeks.
  Will be measured in µM

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Data analysis will be performed in-house.